CLINICAL TRIAL: NCT02620228
Title: INJ-LIVERB-01 Identification of Liver Tumours Using BIP - Biopsy System
Brief Title: Identification of Liver Tumours Using BIP - Biopsy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Injeq Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INJ-LIVERB-01
Record Dates: First submitted 2015-11-20; First posted 2015-12-02 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Liver Biopsy
Keywords: Bioimpedance; Biopsy; Liver tumour; Biopsy needle guidance
MeSH Terms: conditions — Carcinoma, Hepatocellular

ARMS (1):
- BIP Biopsy System (Experimental): Biopsy system that enables real-time bioimpedance measurement from the tip of the biopsy needle.
  Interventions: Device: BIP Biopsy System

INTERVENTIONS:
Device: BIP Biopsy System — BIP Biopsy system is essentially similar as traditional biopsy systems but it enables real-time bioimpedance measurement from the tip of the biopsy needle.

SUMMARY:
This clinical device investigation is conducted by performing liver biopsies using the BIP - Biopsy Tool. The aim is to assess the feasibility of bioimpedance spectroscopy based biopsy tool guidance method and test how well BIP biopsy system is able to distinguish liver tumours from surrounding tissue. In addition, user feedback is obtained to improve the usability of the investigational device. The study does not affect the traditional treatment procedure and only the patients in clinical need for diagnosis by liver biopsy are included on voluntary basis. The invasive products used in actual biopsy operation are designed so that their performance is essentially equal to the currently used biopsy devices, the only difference is the measurement capability of biopsy needle and connection to measurement device.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults undergoing ultrasound-guided core liver biopsy to diagnose liver tumour or other abnormalities
* Identifiable non-tumorous liver tissue along the planned needle injection path.

Exclusion Criteria:

* Inability to give informed consent
* Being under aged
* Being pregnant
* Being high risk patient
* Lack of identifiable non-tumorous liver tissue along the injection path to the tumour location
* Known contraindications to liver biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Difference in mean between measured bioimpedance spectra from tumorous and nontumorous tissue | During liver biopsy (couple of minutes/patient)
  Liver biopsy is performed in traditional way but with biopsy needle that enables bioimpedance measurement from multiple frequencies (spectrum). Tumorous and nontumorous tissue is measured during ultrasound guided biopsy procedure and the tumorous tissue type is verified by histological biopsy sample analysis. The bioimpedance spectra (impedance and phase angle) are compared with each other and differences in means of the spectra calculated. The data analysis is performed offline.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsti Numminen, PhD MD, Principal Investigator — Helsinki University Hospital, Department of Radiology
Locations (1):
- Helsinki University Hospital, Department of Radiology, Helsinki, HUS, Finland